CLINICAL TRIAL: NCT05617443
Title: Comparative Assessment For The Positional Accuracy Of Dental Implants Inserted By Computerized Stackable Surgical Guides Made From Selective Laser Melting And Digital Light Processing Technologies
Brief Title: DLP Versus SLM Stackable Surgical Guide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 535/2022
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-11

CONDITIONS: Accuracy of Stackable Guide
Keywords: implant; stackable guide; 3d printing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- selective laser melting (SLM) CO-Cr metal surgical-guides (Active Comparator)
  Interventions: Device: stackable guide
- digital light processing (DLP) resin surgical-guides (Experimental)
  Interventions: Device: stackable guide

INTERVENTIONS:
Device: stackable guide — different types of stackable guide

SUMMARY:
Purpose; The purpose of this research is to make a comparative estimation for the positional accuracy of dental implants inserted by selective laser melting and digital light processed computerized stackable surgical guides for patients with maxillary terminal dentitions.

Materials and methods; Twenty-four dental implants will be installed in partially edentulous patients who will be applied for treatment of tooth loss and required fixed prosthodontic rehabilitation. Virtually designed prosthetically driven fixation base with its stackable surgical osteotomy guide will be used for bone reduction after tooth extraction and osteotomy preparation respectively. The inserted implants will be divided equally into two groups according to stackable surgical osteotomy guide to either selective laser melting (SLM) CO-Cr metal or digital light processing (DLP) surgical-guides. The final actual implant position will be compared to the preoperative planned position and the deviations will be calculated for coronal deviation, apical deviation in mm, and two angular deviation measurements in degrees.

DETAILED DESCRIPTION:
Preoperative evaluation:

intra-oral and extra-oral examination and medical history for each patient will be recorded to assure that the patient will be eligible for the research.

Written informed consent will be assigned by the patients who will be included in the study.

Preoperative records Polyvinyl siloxane (PVS) impressions for both arches will be made. Also, an interocclusal record will be recorded.

The poured upper and lower cast will be mounted on the articulator and will be scanned using a tabletop scanner (DOF swing, DOF, Korea). the scanned file will be saved in stl format Clinical digital photographs for digital smile design will be used to generate a smile design driven by an individual's face and smile display. As such, it is critical to have at least two portraits representing the lips at rest and another one for a broad smile For each patient, a preoperative cone beam computed tomography (CBCT) scan with the two jaws separated via cotton rolls to separate the volume of interest using a CBCT machine (Scanora 3Dx, Soredex- Finland ) will be taken and saved as Digital Imaging and Communication in Medicine (DICOM) files. The saved STL files will be imported into computer-aided design (CAD) software ( Implastation, prodigident, USA) and superimpose these files to the DICOM files and the JPEG photo files.

Implant and prosthesis planning Virtual tooth setup of the desired prosthetic outcome can be designed to achieve true, restoratively driven implant placement when applied to 3-D surface DICOM data. Performing this virtual wax-up will be done by selecting and importing maxillary teeth from the software library, followed by adjustment of each tooth shape and position according to the patient's occlusion, gender, and smile. The final plan often requires bone reduction to facilitate implant placement and the necessary restorative space for the prosthesis.

A 3-dimensional implant planning using a Software Planning program (Implastation, ProDigident, USA), allows the clinicians to evaluate the osseous tissues concerning the ideal prosthetic position of the virtual waxed-up maxillary teeth. From this information, the sizes and implant receptor sites will be digitally evaluated in all of the necessary views, including cross-sectional, coronal, sagittal, and axial sections followed by virtual placement of the implants.

The stackable guide that will be planned to transfer the virtual plan to the operating field intraorally and consists of 3 components:

1. carrier guide: it takes its support from the remaining dentition and has a foundation base attached to it by locks. its function is to transfer the foundation base to its accurate place in the patient mouth.
2. foundation base: fixed to bone along the whole surgery time by fixation pins and has locks to be attached with subsequent osteotomy guides.
3. osteotomy guide: contains the hole through which the implant drilling will be guided.

The outline of the surgical guide will be determined. and then the thickness and path of insertion. the amount of bone to be reduced will be determined .. a tooth-supported carrier (pin guide) will be designed, it takes its support from the remaining dentition. height of the foundation guide and locations of widely separated 4 anchor pins will be planned so that anchor pins help in achieving the highest degree of surgical accuracy, and then a tooth-supported carrier (pin guide) will be designed, it takes its support from the remaining dentition and accurately replicates the position of the anchor pins for subsequent guides, hence ensuring an accurate replication of the guide position.

With this protocol, teeth removal and bone reduction will be done virtually to provide the available restorative space (from the crest of the bone to the proposed incisal edge position and posterior occlusal plane).

Sleeveless osteotomy guide holes and offset will be designed corresponding to the guided drill kit that will be used(OGS guided kit, oxy implant, Italy) Finally, all guides will be exported as standard triangle language (STL) files and sent to additively manufactured machines.

Grouping:

The inserted implants will be divided equally into two groups according to the stackable surgical osteotomy guide fabrication/printing technique:

First group; in which implants will be placed using selective laser melting (SLM) CO-Cr metal surgical-guides Second group; in which implants will be placed using digital light processing (DLP) resin surgical-guides

Surgical stents fabrication:

For Digital light processing (DLP): DLP printers have a digital projector screen used to flash a single image of each layer on the entire platform at once using curable photopolymer resin. A vat of liquid photopolymer will be exposed to UV light from a digital projector under safelight conditions. The printer (Photon, Anycubic, China) builds the stent one layer at a time by tracing a laser beam on the surface of a vat of printable Resin liquid (SG resin, pro shape, turkey). The process will be repeated, forming another layer on top of the previous layer. This process continues layer by layer until the stent is completed. Printing will be started with a build angle of 45 and the printing thickness on the z-axis was set at 100 microns. After printing, the supports will be removed and the printed stents will be cleaned in an ultrasonic bath with ethyl alcohol for 2 minutes to remove excess resin. Stents will be post-polymerized for 30 minutes using an ultraviolet polymerization unit (bre. Lux power Unit 2, Bredent, Germany).

Regarding Selective Laser Melting (SLM); the STL file will be segmented into cross-sectional layer representations and then exported to a metal laser melting machine (vm120, Vulcan tech, Germany). To fabricate the prototype, this automated printing machine received numerical inputs of the surgical stent design. Sintering of the powder alloy (Starbond easy Pulver 30, Scheftner dental, Germany) to the predesigned guide via high-energy laser beams that traced across a powder bed of densely compacted powdered material, resulting in local melting and fusing of the particles. According to the 3D data fed into the machine, metallic powders will melt together, in a layer-by-layer strategy, creating three-dimensional objects.

Laser spot diameter of 0.08-0.1 mm, sintering speed of 1100-1200 mm/s, a layer thickness of 0.02 mm, and printing angle of 45 degrees, will be considered the parameters of the laser melting machine that will be used for the SLM stent fabrication. SLM stents will be extracted from the base plate and homogenization treatment will be performed at 1150ᵒ C for 30 minutes.

Surgical phase All surgeries will be performed by the same operator under complete aseptic conditions. The patients will be locally anesthetized.

Utilizing the existing dentition to position carrier resin guide to which everything else will be related. Verification of the carrier guide of the pin guide over the teeth will be done.

After verification, the carrier will be securely locked to the foundation metal printed guide and delivered over the teeth. This method allows for the metal foundation guide to be correctly positioned. Four anchor pins will be utilized to stabilize the metal foundation guide (divided equally into anterior and posterior regions bilaterally). An anchoring twist drill will be used with copious irrigation for the preparation of the fixation screw pathway. After that, four anchoring screws will be driven in the anterior and posterior areas After the FG will be secured to the bone, the pin guide will be removed, leaving the maxillary teeth available for extraction. The teeth will be all carefully removed, leaving the remaining alveolus exposed. The outer aspect of the metal FG will be used to determine the amount of bone reduction. Once the alveoloplasty will be completed after the elevation of the palatal flap, a third surgical template which is the stackable osteotomy surgical stent will be positioned and mechanically locked to the top of the FG for guided implant placement.

The osteotomy sites will be prepared, through the planned locations and angulations of the surgical guides, using a sequential series of drills of the OGS Surgical Kit After the last drill, six (NeoBiotech Co., Seoul, Korea) implants will be placed freehand after using drill guides, and tightened manually to 35N/cm. Finally, cover screws will be tightened (10 N/cm) to the implants and the surgical guides were removed. The patients will be instructed to complete the course of antibiotic and anti-inflammatory for 5 days after surgery, to maintain good oral hygiene.

Evaluation After the surgery, patients will be submitted to a CBCT scan using the same parameter as the preoperative scan. And the data of the postoperative scan will be superimposed over the preoperative plan to assess the accuracy of the implant placement using the software (blueskybio 4, BlueSky bio, USA). The final actual implant position will be compared to the preoperatively planned position and the deviations will be calculated for global angel deviation and global linear coronal and apical deviation in mm.

ELIGIBILITY:
Inclusion Criteria:

* well healthy patients
* patients with maxillary terminal dentition

Exclusion Criteria:

* Patients with, systemic disease that might complicate post-operative healing or contribute to bone resorption
* patients with parafunctional habits, poor oral hygiene, limited mouth opening, severe alveolar bone deficiencies,
* patients with uncontrolled diabetes, current irradiation to the head or neck, psychological disorders, or alcohol, tobacco, or drug abuse

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
global angel deviation and global linear coronal and apical deviation in mm. | 1 weekk
  patients will be submitted to a CBCT scan using the same parameter as the preoperative scan. And the data of the postoperative scan will be superimposed over the preoperative plan to assess the accuracy of the implant placement using the software (blueskybio 4, BlueSky bio, USA). The final actual implant position will be compared to the preoperatively planned position and the deviations will be calculated for global angel deviation and global linear coronal and apical deviation in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Hebeshi, Ismailia, Egypt